CLINICAL TRIAL: NCT02036216
Title: Detected the Valuable Characteristic Changes Both in Circulating Cell-free DNA and Primary Tumor in the Patients With Hepatocelluar Carcinoma.
Brief Title: Circulating Cell-free DNA as a Predictive Biomarker for Hepatocelluar Carcinoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: CFD-J14
Record Dates: First submitted 2014-01-07; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma；cell free tumor DNA; Mutation;
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Human plasma；Human blood cells without plasma; HCC tissues (frozen);
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatocellular Carcinoma: The mutation will be found in the DNA samples from the plasma and solid tumor tissues in the patients with HCC.

SUMMARY:
Circulating free cell DNA (cfDNA) is extracellular fragmentation of nucleic acids that occurs both in plasma and serum. This kind of DNA which derived from the apoptotic/necrotic cells or the lysis of circulating tumor cells (CTCs) can be detectedin the patients with a variety of diseases. Emerging evidence suggests that cfDNA from patients exhibits characteristicchanges of tumors, suchas mutations, insertions/deletions, methylations,microsatellite aberrations, and copy number variations, etc. All of these reveal a visible difference between the benign conditions, and thus may be useful in the diagnosis of cancer, identification of targeted therapy, monitor responses to treatments, and early detection of relapse. The purpose for this study is to explore these characteristic changes in the patients withhepatocellular carcinoma (HCC) and expect to guide targeted therapy and identify non-invasive biomarkers of cancer diagnosis and prognosis which can be easily isolated from the circulation.

DETAILED DESCRIPTION:
In cancer, cfDNA can be detected a higher concentration in the circulation because of the necrosis of neoplasm cells with the rapid enlargement and relatively shortage of blood supply. So, identifying tumor-specific genetic and epigenetic changes in cfDNA on this status, such as gene mutations, deletions, methylation alterations and microsatellite alterations, may be more specific for us to diagnose the neoplasms in early phase. This phenomenon also appears in the patients with hepatocellular carcinoma (HCC). Studies have shown that cfDNA level is associated with intrahepatic and extrahepatic metastasis in HCC patients and examined some cfDNAcharacteristic changes, such as p161NK4A, RTL, RASSF1A, LINE-1 and GSTP1. Thus is useful for us to explore the specific cfDNA in HCC. For a high sensitivity and specificity detection, we will use technologiesdeveloped at Stanford Genome Technology Centerto find more characteristic gene mutations, methylation alterations or other changes (3). In this study, we willinvestigate thesecharacteristic changesin cfDNA and primary tumor lesions.

Study arrangement:

Collect the DNA samples from the plasma, blood cells and solid tumor tissues in the patients with HCC.

Detect the DNA sequence from the samples of plasma, blood cells and solid tumor tissues.

Identify cancer specific variations in cfDNA and primary tumor lesions. Date analysis and investigate these characteristic changes. Evaluate the application in early diagnosis, treatment monitoring and prognosis for HCC.

ELIGIBILITY:
Inclusion Criteria:

Age≥18years and ≤80 years; Histologically and cytologically proven Hepatocellular carcinoma Child-Pugh：child A-B Adequate hematological, renal, cardiac and pulmonary functions Tumor in any segment of liver

Exclusion Criteria:

Uncontrolled systemic disease Reject the surgical treatment Metastatic carcinoma Child-Pugh：child C

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The HCC patients who will receive the surgical treatment in Peking Union Medical College Hospital from Jan of 2014 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-06 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
To collect the DNA samples from the plasma, blood cells and solid tumor tissues in the patients with HCC. | three months
  In the first three months in this study, we will collect 5 samples from the plasma, blood cells and primary tumor lesions in the patients with HCC in three stages including preoperative, postoperative (2 weeks) and postoperative (1 month). It is better for us to find the characteristic changes when we make a detailed comparison between the samples in these period. These samples include 5ml plasma, 2ml blood cells without plasma and at least 10mg solid tumor tissues.

SECONDARY OUTCOMES:
Investigate the value characteristic changes from the DNA samples. | three months
  We will prepare the DNA samples from the plasma, blood cells and primary tumor lesions in the patients with HCC in Stanford Genome Technology Center. And then, we will finish DNA sequence in both of them. The DNA sequence which detect from the blood cells will be a normal standard, and thus will be compared with the DNA sequence detect in the samples of plasma and tumor tissues. In this way, we expect to find the common mutations in cfDNA and primary tumor lesions.
Date analysis | two months
  Date analysis will help us to find the changes which have the highest probability in DNA sequence. After that, we will screen these characteristic changes and confirm the sensitive and special mutations which can help us to diagnose the HCC in early phase.
Evaluate the sensitivity and specificity with these changes in HCC | four months
  After we find these valuable characteristic changes in HCC, 50 samples will be detected within these changes. On the basis of the deepen date analysis, we will evaluate the sensitivity and specificity with these changes in HCC.
Early diagnosis, treatment monitoring and prognosis evaluation. | twelve months
  After we complete the evaluation and determine which genetic changes can be used, we will choose 100 patients with HCC and 50 patients who have accepted the surgery treatment in this trial phase. The first 100 patients will be detected these changes before the operation. After that, we expect to establish an evaluation system for early diagnosis in HCC. The postoperative patients will accept the cfDNA detection in the same way with the purpose of estimating the recurrence of the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Yilei Mao, MD, Principal Investigator — PUMCH
Locations (2):
- Stanford Genome Technology Center, Stanford, California, United States
- Department of liver surgery; Peking Union Medical College Hospital；, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Chen K, Zhang H, Zhang LN, Ju SQ, Qi J, Huang DF, Li F, Wei Q, Zhang J. Value of circulating cell-free DNA in diagnosis of hepatocelluar carcinoma. World J Gastroenterol. 2013 May 28;19(20):3143-9. doi: 10.3748/wjg.v19.i20.3143. PMID 23716996
- [Background] Gall TM, Frampton AE, Krell J, Habib NA, Castellano L, Stebbing J, Jiao LR. Cell-free DNA for the detection of pancreatic, liver and upper gastrointestinal cancers: has progress been made? Future Oncol. 2013 Dec;9(12):1861-9. doi: 10.2217/fon.13.152. PMID 24295416
- [Background] Shen P, Wang W, Chi AK, Fan Y, Davis RW, Scharfe C. Multiplex target capture with double-stranded DNA probes. Genome Med. 2013 May 29;5(5):50. doi: 10.1186/gm454. eCollection 2013. PMID 23718862